CLINICAL TRIAL: NCT05901168
Title: Comparison of Acute Responses of Active Video Games and Traditional Exercise Program in Patients With Pulmonary Hypertension
Brief Title: Acute Responses of Active Video Games and Traditional Exercise Program in in Patients With Pulmonary Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Ezgi Ceren Ozcan, Master of Science Student, Dokuz Eylul University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DokuzEU-PAH-001
Record Dates: First submitted 2023-05-03; First posted 2023-06-13 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Hypertension
Keywords: pulmonary hypertension; active video games
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Video Games Intervention (Active Comparator): Active video games intervention will be carried out with a virtual reality system (XBOX360, Microsoft, USA) consisting of a console and sensor.
  Active video games consist of Rally Ball, Rive Rush and Reflex Ridge games.
  Interventions: Other: Active Video Games Intervention
- Traditional Exercise Intervention (Active Comparator): Traditional Exercise Intervention consist of active exercises for the upper extremities, active exercises for the lower extremities, active exercises for the body.
  Interventions: Other: Traditional Exercise Intervention

INTERVENTIONS:
Other: Active Video Games Intervention — Participants will complete active video games in the same order until they fill 20 minutes after the first 5 minutes of warm-up. In addition, during the change between games (lasting approximately 20 seconds), patients will be instructed by a therapist to perform combined exercises to minimize immobility time. These exercises are: elbow flexion and foot flexion, shoulder flexion and unilateral hip extension, and arm abduction and squat exercises that will prevent the patient from cooling down.
  Arms: Active Video Games Intervention
Other: Traditional Exercise Intervention — Active exercises for the upper extremities (without support): Shoulder flexion, Shoulder abduction, Elbow flexion at shoulder 90° flexion.
  Active exercises for the lower extremities: Ankle-foot movements (ankle pumping exercise), heel raise, Knee extension in sitting high, Hip-knee flexion while lying supine
  Body: Bridging, Trunk rotations in sitting
  These exercises will be done in 1 set of 8-10 repetitions.
  It will take about 20 minutes.
  Arms: Traditional Exercise Intervention

SUMMARY:
At least 20 volunteers with a diagnosis of Pulmonary Hypertension in the Department of Cardiology of Dokuz Eylul University and who meet the criteria for follow-up and inclusion will participate in the study. The aim of this study is to examine the acute effects of active video games compared to traditional exercise and the effects on energy expenditure and enjoyment in PH patients. Demographic and clinical information of the participants will be questioned. Active video games and home-based exercise sessions will be held randomly/by the same person with a break of at least 1 day in 1 week, lasting 20 minutes. Heart rate, blood pressure, shortness of breath and oxygen saturation will be measured before and after the sessions. In addition, energy expenditure, heart rate, perceived exertion, shortness of breath and oxygen saturation will be recorded during the sessions. In addition, arterial stiffness will be evaluated with a non-invasive device. At the end of the sessions, whether people like active video games or not will be questioned with a 10-point Likert-type scale.

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) is a progressive disease that can lead to death as a result of right ventricular overload and right heart failure. Early diagnosis and treatment are important. In cardiac catheterization, it is defined as the measurement of mean pulmonary artery pressure above 20 mmHg. Exercise training in Pulmonary Disease has benefits such as improving endothelial dysfunction, muscle blood supply, peripheral O2 extraction, muscle strength, ventilation efficiency, ventricular contractility, reducing adrenergic tone, increasing vagal modulation, and restoring baroreflex arterial sensitivity. There are studies and meta-analyses that show that exercise programs applied under supervision in addition to optimal medical treatment and tailored to the patient have positive effects on functional capacity and quality of life in all Pulmonary Disease groups. Active video games are reported as a useful method to increase adherence to physical exercise routines. Active video games are defined as: playing video games that require intense physical exercise, for exercise purposes, and in which the participant moves large muscle groups in response to cues. It has been reported that active video games that require physical exertion can improve physical activity. Body movements performed in active video games result in varying levels of intensity and energy expenditure. Studies investigating energy expenditure in various age groups have shown that active video games promote physical activity and increase energy expenditure at levels appropriate for moderate to vigorous physical activity. However, the effect of active video games on energy expenditure, attainment of moderate intensity, and acute responses in individuals with Pulmonary Disease compared to conventional exercise has not been clearly investigated. The aim of this study is to examine the acute effects of active video games compared to traditional exercise and the effects on energy expenditure and enjoyment in Pulmonary Disease patients.

Each patient will complete the exercise training and active video game intervention in random order and different days. Active video games intervention will be carried out with a virtual reality system (XBOX360, Microsoft, USA) consisting of a console and sensor. Active video games; will consist of River Rush, Rally Ball and Reflex Ridge games. Traditional-Based Exercise Intervention will consist of active exercises for the upper extremity (without support), active exercises for the lower extremities and body exercises.upper extremity exercises are shoulder flexion, shoulder abduction, elbow flexion at shoulder 90° flexion. Lower extremity exercises are: ankle-foot movements (ankle pumping exercise) heel raise, knee extension in sitting high, hip-knee flexion while lying supine. Body exercises are: bridging andtrunk rotations in sitting. Before and after the sessions; acute responses, vascular responses and enjoyment will be measured. In addition, energy expenditure will be recorded during the sessions.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with PH
* Volunteering
* Being clinically stable
* New York Heart Association 1-3 class
* Have not received physiotherapy in the last 6 months

Exclusion Criteria:

* Presence of unstable angina
* Presence of severe neurological, pulmonary and musculoskeletal disease
* The patient's desire to quit the study
* Playing more than 20 minutes of active video games 3 days a week
* Pregnancy
* Having significant and uncompensated visual and auditory deficiencies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Exercise load end heart rate | Change from baseline to end of 20 minutes of exercise loading
  It will be measured with a pulse oximeter at the end of 20 minutes of exercise loading.
Exercise load end blood pressure | Change from baseline to end of 20 minutes of exercise loading
  It will be measured with a sphygmomanometer at the end of 20 minutes of exercise loading.

SECONDARY OUTCOMES:
Exercise load end perceived effort | Change from baseline to end of 20 minutes of exercise loading
  The degree of perceived effort will be evaluated with the Modified Borg Scale (M.Borg 0-10) at the end of 20 minutes of exercise loading. As the modified borg score of the person increases, the perceived effort will increase.
Exercise load end oxygen saturation | Change from baseline to end of 20 minutes of exercise loading
  Oxygen saturation will be evaluated by pulse oximetry at the end of 20 minutes of exercise loading.
Exercise load end shortness of breath | Change from baseline to end of 20 minutes of exercise loading
  Shortness of breath will be assessed with the Modified Borg Scale(M.Borg 0-10) at the end of 20 minutes of exercise loading after warming up. As the modified borg score of the person increases, the perceived shortness of breath will increase.
Evaluation of energy expenditure | During exercise intervention, average 20 minutes
  Energy expenditure during active video games and traditional exercise will be evaluated using the activity monitor. The activity monitor will be attached to the upper arm. Its accelerometer measures skin temperature, galvanic skin response and heat flux, as well as energy expenditure during movement.
Evaluation of Arterial stiffness | Change from baseline to end of 20 minutes of exercise loading
  Arterial stiffness will be measured with a noninvasive method with the help of the SphygmocorXCEL device, which can automatically measure with the cuff. By means of a transducer, the pressure on the brachial artery will be increased (augmentation index) and carotid-femoral pulse wave velocity (pulse wave velocity) measurements will be made over the artery.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Izmir, Balcova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No